CLINICAL TRIAL: NCT02612454
Title: An Open-Label Extension Study to Assess the Long-Term Safety and Efficacy of Dupilumab in Patients ≥6 Months to <18 Years of Age With Atopic Dermatitis
Brief Title: Study to Assess the Long-term Safety of Dupilumab Administered in Participants ≥6 Months to <18 Years of Age With Atopic Dermatitis (AD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1434; 2015-001396-40 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-23 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Body weight ≥60 kg (Experimental): Administered every two weeks (Q2W)
  Interventions: Drug: Dupilumab
- Body weight 30 kg to <60 kg (Experimental): Administered Q2W
  Interventions: Drug: Dupilumab
- Body weight 15 kg to <30 kg (Experimental): Administered every 4 weeks (Q4W)
  Interventions: Drug: Dupilumab
- Body weight 5 kg to <15 kg (Experimental): Administered Q4W
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Weight-tiered dosing administered subcutaneous (SC)
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
The primary objective of the study is to assess the long-term safety of dupilumab in pediatric participants with AD.

The secondary objectives of the study are:

* To assess the long-term efficacy of dupilumab in pediatric participants with AD
* To assess the trough concentrations of functional dupilumab in serum and the immunogenicity in pediatric participants with AD after re-treatment with dupilumab

Optional Pre-filled Pen (PFP) Sub-Study in pediatric patients ≥2 to <12 years of age with AD

Co-Primary Objectives are:

* To evaluate the pharmacokinetic (PK) of dupilumab PFPs
* To evaluate the safety of dupilumab PFPs

Secondary Objective is:

- To evaluate the immunogenicity of dupilumab PFPs

ELIGIBILITY:
Key Inclusion Criteria:

* Participated in a prior dupilumab study in pediatric participants with AD and adequately completed the visits and assessments required for both the treatment and follow-up periods, as defined in the prior study protocol
* PFP Sub-Study Only:
* Age ≥2 to <12 years at time of screening
* Body weight ≥5 kg and <60 kg at time of screening
* Must have received the same dupilumab dose regimen to be used in the PFP sub-study during the previous 12 weeks in the main OLE study using the prefilled syringe, as defined in the protocol

Key Exclusion Criteria:

* Participants who, during their participation in a prior dupilumab study developed an adverse event (AE) or serious adverse event (SAE) deemed related to study drug which could indicate that continued treatment with study drug may present an unreasonable risk for the patient
* Participants, who during the participation in a prior Dupilumab study, developed an AE that was deemed related to study drug and led to study treatment discontinuation, which in the opinion of the investigator or medical monitor could indicate that continued treatment with study drug may present an unreasonable risk for the patient
* Treatment with an investigational drug, other than dupilumab, within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
* Having used immunosuppressive/immunomodulating drugs within 4 weeks before the baseline visit
* Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit
* Diagnosed active endoparasitic infections or at high risk of these infections
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the participant's participation in the study
* PFP Sub-study Only:
* Poor compliance as defined by having missed 1 or more of the planned last 3 injections in the main OLE study prior to entering the sub-study
* Switched dupilumab doses within the past 12 weeks
* Meet criteria for temporary/permanent discontinuation of study drug at time of screening into PFP sub-study, as defined in the protocol.

Note: Other protocol defined Inclusion / Exclusion criteria may apply

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 880 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment-emergent adverse events (TEAEs) per participant year from baseline through the last study visit | Baseline up to week 272
Number of participants with at least one TEAE per participant year from baseline through the last study visit | Baseline up to week 272
OPTIONAL SUB-STUDY: Pharmacokinetic (PK) of dupilumab: Peak concentration (Cmax) | Up to week 16
  Peak serum concentration after multiple doses of dupilumab administered using the PFP (test) relative to the prefilled syringe (reference)
OPTIONAL SUB-STUDY: PK of dupilumab: Trough concentration (Ctrough) | Up to week 16
  Drug concentration in serum after multiple doses of dupilumab administered using the PFP (test) relative to the prefilled syringe (reference)
OPTIONAL SUB-STUDY: Incidence of TEAEs during the 12-week PFP treatment period and during entire sub-study | Up to week 16
OPTIONAL SUB-STUDY: Incidence of SAEs during the 12-week PFP treatment period and during entire sub-study | Up to week 16

SECONDARY OUTCOMES:
Number of treatment-emergent serious adverse events (SAEs) from baseline through the last study visit | Baseline up to week 272
Incidence of TEAEs of special interest from baseline through the last study visit | Baseline up to week 272
Proportion of participants with an Investigator Global Assessment (IGA) score of 0 or 1 (clear or almost clear) at all in-clinic visits post-baseline | Baseline up to week 272
Proportion of participants with Eczema Area and Severity Index (EASI)-75 (≥75% reduction in EASI from baseline of parent study) response at all in-clinic visits post-baseline | Baseline up to week 272
Change from baseline in EASI score at all in-clinic visits post-baseline | Baseline up to week 272
Percent change from baseline in EASI at all in-clinic visits post-baseline | Baseline up to week 272
Change from baseline in Body Surface Area (BSA) affected by AD (BSA) at all in-clinic visits post-baseline | Baseline up to week 272
Percent change from baseline in SCORing Atopic Dermatitis (SCORAD) at all in-clinic visits post-baseline | Baseline up to week 272
Change from baseline in Children's Dermatology Life Quality Index (CDLQI) for participants ≥4 years of age at all in-clinic visits post-baseline in which the assessments are planned to be performed | Baseline up to week 272
Change from baseline in Infants' Dermatology Quality of Life Index (IDQOL) for participants <4 years of age at all in-clinic visits post-baseline in which the assessments are planned to be performed | Baseline up to week 272
Proportion of responders (defined as participants with IGA 0 or 1) who maintain IGA 0 or 1 during at least 75% of the subsequent* visits during the treatment period | Baseline to week 260
  *Subsequent refers to the visits following the first visit at which IGA 0 or 1 is achieved.
For responders (defined as participants with IGA 0 or 1), median percentage of subsequent* visits during the treatment period, at which IGA 0 or 1 is maintained | Baseline to week 260
  *Subsequent refers to the visits following the first visit at which IGA 0 or 1 is achieved.
Number of AD flares during the study | Baseline to week 272
  AD flares are defined as worsening of the disease that requires escalation/intensification of AD treatment
Annualize event rate of AD flares during the study | Baseline to week 272
  AD flares are defined as worsening of the disease that requires escalation/intensification of AD treatment
Proportion of participants with at least one flare during the study | Baseline to week 272
  AD flares are defined as worsening of the disease that requires escalation/intensification of AD treatment
Proportion of well-controlled weeks | Baseline to week 272
  Well-controlled weeks are those for which participants or parents/caregivers answer "Yes" AND during which no rescue treatments were administered
OPTIONAL SUB-STUDY: Incidence and titer of treatment-emergent anti-drug antibodies (ADA) (PFP Sub-Study) | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (77):
- United States (38):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Gilbert, Arizona
  - Regeneron Investigational Site, Bakersfield, California
  - Regeneron Investigational Site, Long Beach, California
  - Regeneron Investigational Site, Los Angeles, California
  - Regeneron Investigational site, Mission Viejo, California
  - Regeneron Investigational Site, Orange, California
  - Regeneron Investigational Site, Palo Alto, California
  - Regeneron Investigational Site, Rolling Hills Estates, California
  - Regeneron Investigational Site, San Diego, California
  - Regeneron Investigational Site, Centennial, Colorado
  - Regeneron Investigational Site, Washington D.C., District of Columbia
  - Regeneron Investigational Site, Coral Gables, Florida
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Columbus, Georgia
  - Regeneron Investigational Site, Macon, Georgia
  - Regeneron Investigational Site, Sandy Springs, Georgia
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, Skokie, Illinois
  - Regeneron Investigational site, Plainfield, Indiana
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Boston, Massachusetts
  - Regeneron Investigational Site, Ypsilanti, Michigan
  - Regeneron Investigational Site, Plymouth, Minnesota
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Forest Hills, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, Rochester, New York
  - Regeneron Investigational Site, Gahanna, Ohio
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational site, Philadelphia, Pennsylvania
  - Regeneron Investigational Site, Charleston, South Carolina
  - Regeneron Investigational Site, North Charleston, South Carolina
  - Regeneron Investigational Site, Bellaire, Texas
  - Regeneron Investigational Site, Fort Worth, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Investigational Site, Norfolk, Virginia
  - Regeneron Investigational Site, Seattle, Washington
- Canada (9):
  - Regeneron Investigational Site, Calgary, Alberta
  - Regeneron Investigational Site, Surrey, British Columbia
  - Regeneron Investigational Site, Winnipeg, Manitoba
  - Regeneron Investigational Site, Markham, Ontario
  - Regeneron Investigational Site, Ottawa, Ontario
  - Regeneron Investigational Site, Peterborough, Ontario
  - Regeneron Investigational Site, Waterloo, Ontario
  - Regeneron Investigational Site, Windsor, Ontario
  - Regeneron Investigational Site, Montreal, Quebec
- Czechia (3):
  - Regeneron Investigational Site, Kutná Hora
  - Regeneron Investigational Site, Prague
  - Regeneron Investigational Site, Ústí nad Labem
- Germany (8):
  - Regeneron Study Site, Tübingen, Baden-Wurttemberg
  - Regeneron Investigational Site, Frankfurt am Main, Hesse
  - Regeneron Investigational Site, Münster, North Rhine-Westphal
  - Regeneron Investigational Site, Dresden, Saxony
  - Regeneron Investigational Site, Gera
  - Regeneron Investigational Site, Hamburg
  - Regeneron Investigational Site, Munich
  - Regeneron Study Site, München
- Hungary (4):
  - Regeneron Investigational Site, Szolnok, Jász-Nagykun-Szolnok
  - Regeneron Investigational Site, Kaposvár
  - Regeneron Investigational Site, Miskolc
  - Regeneron Investigational Site, Szeged
- Poland (12):
  - Regeneron Investigational Site, Ostrowiec Świętokrzyski, Kielce
  - Regeneron Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Investigational Site, Krakow, Malopolska
  - Regeneron Investigational Site, Katowice, Silesian Voivodeship
  - Regeneron Investigational Site, Bialystok
  - Regeneron Investigational Site, Bydgoszcz
  - Regeneron Investigational Site, Chorzów
  - Regeneron Investigational Site, Gdansk
  - Regeneron Investigational Site, Katowice
  - Regeneron Investigational Site, Krakow
  - Regeneron Investigational Site, Lodz
  - Regeneron Investigational Site, Warsaw
- United Kingdom (3):
  - Regeneron Investigational Site, London, Greater London
  - Regeneron Investigational Site, Manchester, Lancashire
  - Regeneron Investigational Site, Sheffield, South Yorkshire

REFERENCES:
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Paller AS, Siegfried EC, Simpson EL, Cork MJ, Sidbury R, Chen IH, Khokhar FA, Xiao J, Dubost-Brama A, Bansal A. Dupilumab Safety and Efficacy up to 1 Year in Children Aged 6 Months to 5 Years with Atopic Dermatitis: Results from a Phase 3 Open-Label Extension Study. Am J Clin Dermatol. 2024 Jul;25(4):655-668. doi: 10.1007/s40257-024-00859-y. Epub 2024 May 14. PMID 38743155
- [Derived] Cork MJ, Thaci D, Eichenfield LF, Arkwright PD, Chen Z, Thomas RB, Kosloski MP, Dubost-Brama A, Prescilla R, Bansal A, Levit NA. Dupilumab Safety and Efficacy in a Phase III Open-Label Extension Trial in Children 6-11 Years of Age with Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2023 Nov;13(11):2697-2719. doi: 10.1007/s13555-023-01016-9. Epub 2023 Sep 26. PMID 37750994
- [Derived] Blauvelt A, Guttman-Yassky E, Paller AS, Simpson EL, Cork MJ, Weisman J, Browning J, Soong W, Sun X, Chen Z, Kosloski MP, Kamal MA, Delevry D, Chuang CC, O'Malley JT, Bansal A. Long-Term Efficacy and Safety of Dupilumab in Adolescents with Moderate-to-Severe Atopic Dermatitis: Results Through Week 52 from a Phase III Open-Label Extension Trial (LIBERTY AD PED-OLE). Am J Clin Dermatol. 2022 May;23(3):365-383. doi: 10.1007/s40257-022-00683-2. Epub 2022 May 14. PMID 35567671
- [Derived] Paller AS, Tan JKL, Bagel J, Rossi AB, Shumel B, Zhang H, Abramova A. IGAxBSA composite for assessing disease severity and response in patients with atopic dermatitis. Br J Dermatol. 2022 Mar;186(3):496-507. doi: 10.1111/bjd.20872. Epub 2022 Feb 25. PMID 34726270
- [Derived] Bansal A, Simpson EL, Paller AS, Siegfried EC, Blauvelt A, de Bruin-Weller M, Corren J, Sher L, Guttman-Yassky E, Chen Z, Daizadeh N, Kamal MA, Shumel B, Mina-Osorio P, Mannent L, Patel N, Graham NMH, Khokhar FA, Ardeleanu M. Conjunctivitis in Dupilumab Clinical Trials for Adolescents with Atopic Dermatitis or Asthma. Am J Clin Dermatol. 2021 Jan;22(1):101-115. doi: 10.1007/s40257-020-00577-1. PMID 33481203